CLINICAL TRIAL: NCT01536392
Title: Oral Ondansetron Versus Transdermal Granisetron (Sancuso) for Women With Cervical, Endometrial or Vaginal Cancer Receiving Pelvic Chemoradiation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sancuso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-1107; NCI-2012-00221 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Cancer of the Cervix
Keywords: Cancer of the Cervix; Anti-emetic therapy; Granisetron; Transdermal patch; Ondansetron; Zofran; Questionnaires; Surveys; Study Drug Diary; Nausea and Vomiting
MeSH Terms: conditions — Uterine Cervical Neoplasms; Nausea; Vomiting | interventions — Granisetron; Ondansetron; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Granisetron (Experimental): Group A: 34.3 mg of granisetron formulated in transdermal patch replaced every 7 days. Transdermal patch placed/replaced prior to the intravenous (IV) infusion of cisplatin. At cycle 1, participants receive IV granisetron prior to IV cisplatin and prior to administration of transdermal patch.
  Interventions: Drug: Granisetron; Behavioral: Questionnaires; Behavioral: Study Drug Diary
- Ondansetron (Experimental): Group B: 8 mg of ondansetron orally thrice daily starting with cisplatin administration and continued for 72 hours after chemotherapy infusion.
  Interventions: Drug: Ondansetron; Behavioral: Questionnaires; Behavioral: Study Drug Diary

INTERVENTIONS:
Drug: Granisetron — 34.3 mg of granisetron formulated in a transdermal patch replaced every 7 days. At cycle 1, participants receive granisetron by vein prior to IV cisplatin and prior to administration of transdermal patch.
  Arms: Granisetron
Drug: Ondansetron — 8 mg of ondansetron by mouth three times a day starting with cisplatin administration and continued for 72 hours after chemotherapy infusion.
  Other Names: Zofran
  Arms: Ondansetron
Behavioral: Questionnaires — Completion of 3 questionnaires at study visits taking about 5 minutes each time.
  Other Names: Surveys
Behavioral: Study Drug Diary — Study drug diary to record times that study drugs taken, and to record any nausea or vomiting experienced.

SUMMARY:
The goal of this clinical research study is to compare granisetron (when given through a patch) to ondansetron (when taken by mouth) for reducing nausea and vomiting in women with cervical, endometrial, or vaginal cancer having chemoradiation.

Granisetron and ondansetron are designed to help reduce nausea and vomiting.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, and you are among the first 40 participants, you will have an equal chance of being in either group. If you enroll after that, you will have a higher chance (51%-100%) of being assigned to the group that had better results.

* If you are in Group 1, you will receive granisetron by patch.
* If you are in Group 2, you will receive ondansetron by mouth.

Study Drug Administration:

If you are in Group 1, you will receive ondansetron by vein at your first visit only, which is standard of care. Then, you will receive cisplatin by vein over about 1 hour as part of the chemoradiation. A granisetron patch will then be placed on your skin before the chemotherapy . The patch will be replaced every 7 days before the chemotherapy.

If you are in Group 2, you will receive ondansetron by vein before cisplatin. Then, you will receive cisplatin by vein over about 1 hour. Then you will take ondansetron by mouth with a cup of water (8 ounces) 3 times a day for 3 days. Ondansetron is a tablet that you can take with or without food and is best taken at least 30 minutes before eating.

Both groups will be given a study drug diary to record the times that you take the study drugs. You will also record any nausea or vomiting that you may have. You should bring the diary to each study visit. You should also bring your study drug bottles/packages to each study visit.

Study Visits:

The visits for this study will be at the same time as your chemoradiation therapy visits over 5 weeks.

You will complete 3 questionnaires at your study visits and then again 1 week after the last chemotherapy. The last questionnaires will be completed by phone. The questionnaires ask about how easy or difficult it is to use your assigned study drug, your level of nausea and vomiting, and your quality of life. It should take about 5 minutes to complete these questionnaires each time.

Length of Treatment:

You may continue using the study drug up to 5 weeks during your chemoradiation treatment. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over when you have completed 5 weeks of chemoradiation treatments.

This is an investigational study. Both granisetron and ondansetron are FDA approved and commercially available for the treatment of nausea and vomiting. It is investigational to compare these drugs administered in different ways.

Up to 150 patients will take part in this study. Up to 120 participants will take part at MD Anderson. Up to 30 will be enrolled at the Harris Health System.

ELIGIBILITY:
Inclusion Criteria:

1. Women with cervical, endometrial or vaginal cancer dispositioned to receive primary or postoperative adjuvant pelvic radiation therapy with concurrent cisplatin administration.
2. Women must be at least 18 years of age.
3. Women must be able to read English or Spanish at a sixth grade level.
4. Women with childbearing potential must have a negative pregnancy test within 1 week of starting chemoradiation therapy.

Exclusion Criteria:

1. Women with cervical, endometrial or vaginal cancer who are receiving chemotherapy and/or radiation therapy for recurrent disease.
2. Women with cervical, endometrial, or vaginal cancer who are receiving extended field radiation therapy.
3. Women with cervical, endometrial or vaginal cancer who are receiving chemotherapy and/or radiation therapy in a palliative setting.
4. Women with cervical, endometrial, or vaginal cancer who have already received their first dose of chemotherapy or radiation for more than 7 days prior to starting chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M. Frumovitz, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 2012 until June 2016. All the recruitment was done in a medical clinic setting.
Pre-assignment Details: 76 participants signed consent, 1 participant did not receive treatment due to the study closure.
Groups:
- Arm 1: Transdermal Granisetron: 8 mg ondansetron given IV prior to Cycle 1 of Cisplatin then 34.3 mg granisetron patch applied and then reapplied every 7 days prior to Cycles 2-5 of Cisplatin.
- Arm 2: Oral Ondansetron: 8 mg ondansetron given IV prior to Cycles 1-5 then 8 mg oral ondansetron every 8 hours for 72 hours following each Cisplatin and PRN in-between cycles.
Period: Overall Study
Arm/Group | Arm 1: Transdermal Granisetron | Arm 2: Oral Ondansetron
Started | 41 | 34
Completed | 28 | 19
Not Completed | 13 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Non Compliance | 3 | 4
Not completed — Completed therapy early | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Transdermal Granisetron | Arm 2: Oral Ondansetron | Total
Number analyzed (Participants) | 41 | 34 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 31 | 68
  >=65 years | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: Years] | 45 [21 to 80] | 51 [30 to 86] | 49 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 34 | 75
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 33 | 29 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 34 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response Rate to Anti-Emetic Therapy Days 4-7 Each Chemotherapy Cycle
Description: Response defined as no emetic or retching episodes and no rescue medication use during late onset phase (4-7 days post-chemotherapy) measured each cycle. Responses tabulated to 4 items of Morisky Medication Adherence measure for each treatment group by cycle of therapy. Elements summarized of Morrow Assessment of Nausea and Emesis and for pill counts/compliance for each treatment group by cycle of therapy. Descriptive statistics summarize total scores for Osoba Module, used to measure effect of nausea and vomiting on quality of life, for each treatment group by cycle of therapy. Osoba Nausea and Emesis Module; higher scores indicate worse quality of life. Morisky Medication Adherence Scale. Higher scores indicate higher compliance. Morisky Medication Adherence Scale is Yes=0 and No=1 , zero is the lowest level of medication adherence, and 4 is the highest level of medication adherence.
Time Frame: Baseline, up to 7 days post-chemotherapy, through 5 cycles of chemotherapy measured each cycle, an average of 6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Transdermal Granisetron | Arm 2: Oral Ondansetron
Number analyzed (Participants) | 41 | 34
percentage of participants | 49.8 [35.2 to 64.3] | 39.7 [24.4 to 56.1]

2. Secondary Outcome: Percentage of Participants With Response Rate to Anti Emetic Therapy 0-24 Hours Each Chemotherapy Cycle
Description: The response rates to anti-emetic therapy (no emetic or retching episodes and no rescue medication use) in the acute (0-24 hours) phase. Responses tabulated to 4 items of Morisky Medication Adherence measure for each treatment group by cycle of therapy. Elements summarized of Morrow Assessment of Nausea and Emesis and for pill counts/compliance for each treatment group by cycle of therapy. Descriptive statistics summarize total scores for Osoba Module, used to measure effect of nausea and vomiting on quality of life, for each treatment group by cycle of therapy. Osoba Nausea and Emesis Module; higher scores indicate worse quality of life. Morisky Medication Adherence Scale. Higher scores indicate higher compliance. Morisky Medication Adherence Scale is Yes=0 and No=1 , zero is the lowest level of medication adherence, and 4 is the highest level of medication adherence.
Time Frame: Baseline, up to 24 hours post-chemotherapy, through 5 cycles of chemotherapy measured each cycle, an average of 6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Transdermal Granisetron | Arm 2: Oral Ondansetron
Number analyzed (Participants) | 41 | 34
percentage of participants | 49.8 [35.2 to 64.3] | 39.7 [24.4 to 56.1]

ADVERSE EVENTS:
Time Frame: Baseline through 7 days for each chemotherapy cycle, an average of 6 weeks
Arm/Group | Arm 1: Transdermal Granisetron | Arm 2: Oral Ondansetron
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/34
Other Adverse Events (participants affected / at risk) | 15/41 | 12/34
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Transdermal Granisetron (N=41) | Arm 2: Oral Ondansetron (N=34)
Constipation (Gastrointestinal disorders) | 8 | 6
Diarrhea (Gastrointestinal disorders) | 9 | 3
Nausea (Gastrointestinal disorders) | 15 | 12
Fatigue (General disorders) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT01536392/Prot_SAP_000.pdf